CLINICAL TRIAL: NCT05656560
Title: Reducing High Risk Polypharmacy Using Behavioral Economics Through Electronic Health Records
Brief Title: Reducing High-Risk Geriatric Polypharmacy Via EHR Nudges R01 Trial
Acronym: HRPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Pittsburgh Medical Center (Other); University of Southern California (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Professor; Director, Center for Primary Care Innovation, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00213231; R01AG070054 (NIH)
Record Dates: First submitted 2022-11-17; First posted 2022-12-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Polypharmacy
Keywords: clinical decision support; electronic health record; behavioral economics; high-risk geriatric polypharmacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinician education only (Other): Online clinician education
  Interventions: Other: Clinician education
- Commitment nudge (Experimental): The commitment nudge will be an EHR alert that is triggered when a clinician renews or orders a qualifying medication in any Epic encounter (including non-face-to-face encounters) for a patient aged 65 or greater who meets criteria for high-risk polypharmacy. When triggered, the commitment nudge will offer the clinician a choice option that sets a reminder to discuss polypharmacy at the patient's next visit date.
  Interventions: Behavioral: Clinical decision support (CDS)-Commitment nudge; Other: Clinician education
- Justification nudge (Experimental): The justification nudge will be an EHR alert triggered for patients with high-risk polypharmacy when a clinician begins to renew or newly prescribe a medication that causes a high-risk criterion to be fulfilled (i.e., a medication meeting causing 1 of the 7 high-risk polypharmacy criteria/primary study measures to be met). This alert will inform the clinician of the high-risk nature of the prescription and request a free-text justification for starting or renewing the medication. This written justification will appear in the EHR in a section of that encounter that other EHR users can see.
  Interventions: Other: Clinician education; Behavioral: Clinical decision support (CDS)-Justification nudge
- Commitment nudge + Justification nudge (Experimental): This study arm will receive both the commitment nudge and the justification nudge.
  Interventions: Behavioral: Clinical decision support (CDS)-Commitment nudge; Other: Clinician education; Behavioral: Clinical decision support (CDS)-Justification nudge

INTERVENTIONS:
Behavioral: Clinical decision support (CDS)-Commitment nudge — EHR clinical decision support alerts-clinician commitment to discuss high risk polypharmacy
  Other Names: Commitment nudge
  Arms: Commitment nudge; Commitment nudge + Justification nudge
Other: Clinician education — Brief, online education module for primary care clinicians
Behavioral: Clinical decision support (CDS)-Justification nudge — EHR clinical decision support alerts-clinician rational for high risk polypharmacy
  Other Names: Justification nudge
  Arms: Commitment nudge + Justification nudge; Justification nudge

SUMMARY:
High-risk polypharmacy is common among older adults in the United States, is particularly dangerous for individuals with dementia or cognitive impairment, and is associated with harms such as adverse drug reactions, falls, and higher costs of care. This project aims to test in a pragmatic clinic-randomized controlled trial two electronic health record-based behavioral economic nudges to help clinicians reduce high-risk polypharmacy among their older adult patients and in the subgroup with dementia or cognitive impairment.

The main questions this trial aims to answer are:

Aim 1: To evaluate the effects of an EHR-based commitment nudge, a justification nudge, and the combination of both nudges on a composite measure of high-risk polypharmacy via a pragmatic randomized controlled trial. The investigators will use cluster randomization in which primary care clinics are randomized to receive 0, 1, or 2 nudges using a factorial design. The nudges will run for 18 months, followed by 12 months of observation to assess persistence of effects.

Aim 2: To qualitatively and quantitatively assess clinician experiences with the EHR-based nudges, including their acceptability and effects on workflow. At the conclusion of the intervention period, the investigators will perform semi-structured interviews and field a clinician survey.

ELIGIBILITY:
Inclusion Criteria:

* Northwestern Medicine or UPMC primary care clinic: Internal Medicine, Family Medicine, or General Practice or Geriatrics

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of HRPP with any (1 or more) of the 7 measures of high risk polypharmacy. (Composite measure) | 18 months
  The composite of the 7 high-risk polypharmacy measures (Secondary outcomes #6-12)

SECONDARY OUTCOMES:
The rate of Emergency Department visits per patient -all cause | 18 months
  Denominator: All older adults with HRPP. Numerator: Patients with an emergency department encounter during the look back period.
The rate of Emergency Department visits per patient-Adverse drug event (ADE)-specific | 18 months
  Denominator: All older adults with HRPP. Numerator: Patients with an emergency department encounter for ADE during the look back period.
The rate of hospital admissions per patient-all cause | 18 months
  Denominator: All older adults with HRPP. Numerator: Patients with an inpatient admission for any reason during the look back period.
The rate of hospital admissions per patient-ADE-specific | 18 months
  Denominator: All older adults with HRPP. Numerator: Patients with an inpatient admission for ADE during the look back period.
The percentage of HRPP patients with a fall condition-drug interaction | 18 months
  Denominator: All older adult patients with HRPP with a fall marker. Numerator: Patients with an active eligible fall risk medication on medication list.
The percentage of HRPP patients with a fall drug-drug interaction | 18 months
  Denominator: All older adult patients with HRPP. Numerator: Patients with greater than or equal to 3 active eligible fall risk medications.
The percentage of HRPP patients with Heart failure-NSAID interaction | 18 months
  Denominator: All older adult patients with HRPP with a CHF marker. Numerator: Patients with an active eligible NSAID medication.
The percentage of HRPP patients with Heart Failure-thiazolidinedione interaction | 18 months
  Denominator: All older adults with HRPP with a CHF marker. Numerator: Patients with an active eligible thiazolidinedione medication.
The percentage of HRPP patients with Heart failure with reduced ejection fraction- non-dihydropyridine calcium channel blocker interaction | 18 months
  Denominator: All older adults with HRPP with CHFlowEF marker. Numerator: Patients with an active eligible calcium channel blocker medication.
The percentage of HRPP patients with CKD-glyburide/glimepiride interaction | 18 months
  Denominator: All older adults with HRPP with most-recent eGFR <60. Numerator: Patients with an active eligible glyburide-containing medication.
The percentage of HRPP patients with CKD-NSAID interaction | 18 months
  Denominator: All older adults with HRPP with most-recent eGFR < 30. Numerator: Patients with an active eligible NSAID medication.

OTHER OUTCOMES:
The percentage of HRPP patients with a hospitalization or emergency department (ED) visit for seizure. | 18 months
  Safety measure for discontinuing or reducing benzodiazepines and anticonvulsants
The percentage of HRPP patients with a hospitalization or ED visit for pain. | 18 months
  Safety measure for discontinuing or reducing tricyclic antidepressants, gabapentinoids, serotonin and norepinephrine reuptake inhibitors, opioids, and NSAIDs
The percentage of HRPP patients with a hospitalization or ED visit for depression or suicidality | 18 months
  Safety measure for discontinuing or reducing tricyclic antidepressants, serotonin and norepinephrine reuptake inhibitors and selective serotonin reuptake inhibitors
The percentage of HRPP patients with a hospitalization or ED visit for anxiety. | 18 months
  Safety measure for discontinuing or reducing benzodiazepines, serotonin and norepinephrine reuptake inhibitors and selective serotonin reuptake inhibitors
The percentage of HRPP patients with a hospitalization or ED visit for sedative withdrawal. | 18 months
  Safety measure for discontinuing or reducing benzodiazepines and Z-drugs (GABA receptor modulators)
The percentage of HRPP patients with a hospitalization or ED visit for opioid withdrawal. | 18 months
  Safety measure for discontinuing or reducing opioids
The percentage of HRPP patients with a hospitalization or ED visit for behavioral disturbance in dementia or psychosis. | 18 months
  Safety measure for discontinuing or reducing antipsychotics
The percentage of HRPP patients with a hospitalization or ED visit for hyperglycemia. | 18 months
  Safety measure for discontinuing or reducing glyburide, glimepiride, and thiazolidinediones
The percentage of HRPP patients with a hospitalization or ED visit for tachycardia (other than ventricular) or hypertensive emergency. | 18 months
  Safety measure for discontinuing or reducing non-dihydropyridine calcium channel blockers

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern Medicine, Chicago, Illinois
  - UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05656560/SAP_000.pdf